CLINICAL TRIAL: NCT06042361
Title: Enhancing Equity in Smoke-free Housing: Evidence-based Strategies to Support Implementation in Permanent Supportive Housing (PSH) Communities
Brief Title: Enhancing Equity in Smoke-free Housing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Vaughan Rees, Director, Center for Global Tobacco Control, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB23-0415
Record Dates: First submitted 2023-07-27; First posted 2023-09-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Tobacco Use Disorder; Second Hand Tobacco Smoke
Keywords: tobacco; second hand tobacco smoke; tobacco cessation; smokefree housing
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Two-phased approach: formative first phase, testing second phase. Enrollment based on residential property clusters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): All participants will receive the intervention of the Smokefree Implementation Framework and Toolkit
  Interventions: Behavioral: Smokefree Implementation Framework and Toolkit

INTERVENTIONS:
Behavioral: Smokefree Implementation Framework and Toolkit — Framework and toolkit that includes "Implementation Guide", "Action Plan", and "Implementation Checklist" that supports the needs of Permanent Supportive Housing communities.

SUMMARY:
The goal of this clinical trial is to learn about the acceptability, feasibility, and effectiveness of smoke-free housing policy implementation in Permanent Supportive Housing communities. The main objective of this study is to identify and refine adaptations for a smoke-free housing implementation framework that incorporates behavioral health support and meets the needs of residents living in Permanent Supportive Housing.

DETAILED DESCRIPTION:
The study aims are:

Aim 1): Identify adaptations for a smokefree housing implementation framework and identify opportunities to integrate these adaptations with ongoing behavioral health support, to meet the needs of residents living in Permanent Supportive Housing (PSH) (Phase 1).

Aim 2): The research team will pilot test the adapted implementation framework, including an implementation toolkit, to assess the acceptability, feasibility and effectiveness of the primary intervention provided to Property Managers (Phase 2).

Aim 3): Based on a synthesis of qualitative and quantitative evidence, the research team will further refine the smokefree implementation framework and toolkit, comprising modified versions of the "Implementation Guide", "Action Plan" and "Implementation Checklist", to support future needs of Permanent Supportive Housing communities (Phase 3).

The research team seeks to use the opportunity provided by smokefree housing implementation to minimize indoor smoking and encourage smoking cessation, and thus help move communities with a history of profound health disparities towards a more equitable, tobacco-free future. The impact of this project will be evident not only among smokers, but also non-smokers, children and the elderly who share residential communities with people supported by PSH programs.

If successful, the results of this work will be used to promote broader and more effective use of the smokefree PSH implementation framework in federally-assisted public and affordable housing communities nationally.

ELIGIBILITY:
The study setting is 6 affordable housing communities that include Permanent Supportive Housing (PSH) in Massachusetts, Maryland and New York (USA).

Inclusion Criteria:

* Adult residents of the six affordable housing communities who smoke or do not smoke tobacco, who receive or do not receive Permanent Supportive Housing services, and can complete a survey in English or Spanish.
* Adult residents of the six affordable housing communities who smoke or do not smoke tobacco, who receive or do not receive Permanent Supportive Housing services, and can participate in a focus group discussion in English.
* Property Managers (or their designated appointees) of the six affordable housing communities where the research will be conducted and able to receive the intervention and participate in the qualitative interviews in English.
* Caseworkers who are dedicated health workers who provide behavioral health support (mental health and substance use support interventions) to residents at each of the six properties and who can receive the intervention and participate in the qualitative interviews in English.

Exclusion Criteria:

* Those unable to speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Pre-intervention through 6 months post intervention
  The Smokefree Implementation Framework and Toolkit is acceptable to implement in Permanent Supportive Housing communities. Measured using 4-items from the AIM.
Feasibility of Intervention Measure (FIM) | Pre-intervention through 6 months post intervention
  The Smokefree Implementation Framework and Toolkit is feasible to implement in Permanent Supportive Housing communities. Measured using 4-items from the FIM.

SECONDARY OUTCOMES:
Ambient second-hand smoke in common indoor areas | Pre-intervention through 6 months post intervention
  Monitored using passive nicotine dosimetry monitors placed in common areas
Residents' self-reported exposure to secondhand smoke | Pre-intervention through 6 months post intervention
  Self-reported exposure to secondhand smoke (smell or sight) in the home or around the property, will be assessed with two questions in survey form.
Behavior of residents who smoke | Pre-intervention through 6 months post intervention
  Self-reported behavior of smoking (cigarettes/day in the past 30 days) of residents who smoke

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan Rees, PhD, Principal Investigator — Harvard University School of Public Health
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No